CLINICAL TRIAL: NCT00123188
Title: Development of a Screening Test for Endometrial Hyperplasia in an At Risk Cohort
Brief Title: Ultrasound and Endometrial Hyperplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: enrollment of participants has halted prematurely; difficulty with recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Center for Research on Women and Health (Unknown)
Responsible Party: Principal Investigator, Richard S. Legro, M.D., Professor, Obstetrics and Gynecology and Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20175
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: Endometrial Hyperplasia
MeSH Terms: conditions — Endometrial Hyperplasia | interventions — High-Energy Shock Waves; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasound and Biopsy (Experimental): Transvaginal Ultrasound and Endometrial Biopsy
  Interventions: Procedure: Ultrasound and Biopsy

INTERVENTIONS:
Procedure: Ultrasound and Biopsy — Transvaginal ultrasound and Endometrial Biopsy

SUMMARY:
The investigators hypothesize that endometrial thickness will be a significant predictor of endometrial hyperplasia in a postmenopausal female population with metabolic syndrome: diabetes and/or insulin resistance, hypertension, and obesity.

DETAILED DESCRIPTION:
The objective is to identify the utility of ultrasound as a screening test for endometrial hyperplasia and cancer in an "at risk" cohort. Endometrial carcinoma is an understudied cancer. This study will provide benefit regardless of its outcome, because it will be the first prospectively designed screening trial in an asymptomatic population.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal obese subjects, who have diabetes or a prediabetic state, or hypertension

Exclusion Criteria:

* Women who have had a hysterectomy

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-04; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Endometrial Hyperplasia | End of study
  A transvaginal ultrasound of the endometrium will be performed to obtain measures of the anteroposterior endometrial thickness (in the sagittal plane), the dimensions of the endometrial cavity (thickness, length and width), and the appearance of the endometrium in addition to uterine and ovarian measures. Endometrial thickness will be a significant predictor of endometrial hyperplasia in a postmenopausal female population with the metabolic syndrome: diabetes and/or insulin resistance, hypertension, and obesity.

SECONDARY OUTCOMES:
Endometrial Cancer | End of study
  All women will then undergo an endometrial biopsy. The pipelle has been shown to be an accurate method of diagnosing endometrial cancer comparable to a full dilatation and curettage of the uterus. We believe it is important to perform a biopsy even in women with a thin endometrial stripe (<5mm), as it will be important for determining the specificity and negative predictive value of both ultrasound and any serum screening strategy we devise.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Legro, M.D., Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey, Hershey, Pennsylvania, United States